CLINICAL TRIAL: NCT01026753
Title: Innovative Tools to Improve Colorectal Cancer Screening Rates in Manitoba
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CancerCare Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Alan Katz, Head of Family Medicine Research, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H2009:312
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; screening; fecal occult blood test; randomized control trial; primary care oncology; web site; provincial health contact center
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOBT by laboratory requisition or directly by PCP (No Intervention): The family physician indicates fecal occult blood test on the patient's laboratory requisition (i.e. the patient receives the fecal occult blood test at the lab) or provides the patient with an FOBT kit.
- FOBT by lab req. or directly from PCP + study magnet (Experimental): The family physician indicates fecal occult blood test on the patient's laboratory requisition (i.e. the patient receives the fecal occult blood test at the lab) or provides the patient with an FOBT kit. The family physician provides each patient with a study magnet containing a PHCC telephone number and study specific website address.
  Interventions: Behavioral: Refrigerator Magnet

INTERVENTIONS:
Behavioral: Refrigerator Magnet — The refrigerator magnet contains a telephone number for a Provincial Health Contact Centre and a URL for a colorectal cancer Website that patients can access to learn more about colorectal cancer, screening and the fecal occult blood test. Patients can also have their questions answered.
  Arms: FOBT by lab req. or directly from PCP + study magnet

SUMMARY:
The primary purpose of the study is to investigate the efficacy and effectiveness of a community-based nurse managed telephone support line (Provincial Health Contact Center; PHCC) and Colorectal Cancer Information and Screening Website in supporting Primary Care Providers (PCP) from Winnipeg, Manitoba (Canada) in their efforts to improve colorectal cancer (CRC) screening Fecal Occult Blood Test (FOBT) compliance in average risk men and women 50-74 years of age. Secondary outcomes of the study involve documenting and investigating common patient questions and comments about CRC and the FOBT during their PHCC communication(s)/Website visits as well as procuring feedback from PCP and patients related to their experiences with the study protocol (PCP), FOBT (patients) and PHCC/website (patients).

DETAILED DESCRIPTION:
Primary care providers (PCP) will be recruited within the Winnipeg Regional Health Authority (WRHA) community areas of St. James Assiniboia, Assiniboine South, Downtown, River Heights, Fort Garry, St. Vital and St. Boniface. The first step in recruiting PCP within the WRHA will involve a pre-collaboration call to PCP/clinics to make them aware that the study coordinator will be dropping off a a PCP Collaboration Letter that briefly outlines the proposed research study and requests the participation of PCP. The letter will inquire as to whether the PCP/clinic would be interested in collaborating on the study as well as the best date, time and method of contacting the office. Based on this information, the study coordinator will contact each clinic in the preferred manner to set a date and time to determine their interest in study collaboration and, if so, to set a date and time for a site visit to discuss the study protocol and PCP/clinic involvement and responsibilities.

Once a PCP/clinic has agreed to collaborate on the study, a PCP/Clinic Characterization Form will be completed by the study coordinator. The purpose of this form is to document the routine standard of care provided by each PCP in regards to CRC screening practices with the FOBT and to ensure minimal obtrusiveness of the study protocol in the daily functioning of the PCP/clinic. It is believed that, in Winnipeg, two standard methods of having patients complete an FOBT exist; laboratory requisition filled out by the PCP or direct distribution of the FOBT kit by the PCP to the patient. By filling out the PCP/Clinic Characterization Form, the preferred method of FOBT screening by each PCP/clinic will be documented. This factor will be taken into account as a covariate in the statistical analysis of the data. All PCP within a medical clinic will be randomly allocated to one of two study groups (control or intervention). In the case of medical clinics where there are sub-groupings of PCP/staff that function as a single/separate unit/entity, each sub-group of PCPs will be randomized separately. The objective of customizing this portion of the study protocol to each PCP/clinic is to optimize collaboration with PCPs as well as simulate "real world" PCP practices resulting in evidence-based findings that are able to be integrated into practice.

Collaborating PCP/clinics will be randomly allocated into providing their average risk male and female patients (50-74 years) with either the control or the intervention protocol for FOBT screening for CRC. As there is one type of control group and one study intervention (provision of a magnet with contact information for a Provincial Health Contact Center (PHCC) and Colorectal Cancer Information and FOBT Screening Website) there are a total of two study groups: (1) FOBT recommendation based on usual PCP practice, and (2) FOBT recommendation based on usual PCP practice + magnet. Once a PCP/Clinic is randomized into a group, all their patients will participate in that study group.

Upon arrival for their periodic health examination (PHE) appointment, eligible patients in all study groups will be asked by a front desk clinic support staff employee to complete an In-Clinic Patient Survey/Consent Form related to their exposure to Provincial CRC Screening initiatives (CancerCare Manitoba; ColonCheck) and whether they have completed an FOBT in conjunction with the CancerCare Manitoba Screening Program in the last two years.

During their PHE, the PCP will determine patient eligibility according to the criteria outlined by the study coordinator during the site visit. PCPs in the control group will provide patients with a laboratory requisition indicating an FOBT or directly provide the FOBT kit to patients. Those patients who have a lab requisition indicating FOBT will receive the FOBT kit from the laboratory. PCP in the control and intervention groups will be provided with Patient Tracking Forms (one per patient) on which the PCP will indicate the patient name and date of FOBT requisition/distribution. Each Patient Tracking Form will have a removable sticker with a unique patient study identification number. The PCP will remove the sticker from the Patient Tracking Form and place it on the patient's In-Clinic Survey which will allow researchers to link the data. Study identification numbers that will facilitate patient tracking as well as allow the study coordinator to determine for each PCP/clinic, the number of patients requested by the PCP/clinic to complete an FOBT. It will also facilitate tracking patients that complete their FOBT. The study coordinator will follow-up with PCP/clinic support staff to determine the patients completing their FOBT. Patients are given four months in which to complete their FOBT. After this time, if the FOBT is not completed, they will be assigned an incomplete according to the intention to treat model. In this way, personal health identification is protected. The study coordinator will contact the PCP/clinics regularly for Patient Tracking Form updates and to foster collaborative relationships between researchers and PCP.

PCP/clinics allocated to the intervention groups will be utilize the same Patient Tracking Forms as described above. Each of the Patient Tracking Form sheets will have a sequentially numbered study magnet attached that the PCP will provide to their patient. The refrigerator magnet contains a study specific PHCC telephone number and Website address as well as a brief message about the importance of the FOBT in early detection of CRC.

The sheets of sequential study identification numbers and the Patient Tracking Forms will facilitate determining the number of patients for which an FOBT was requested and the number of patients provided with a magnet. Patients provided with a magnet will use the number assigned to their magnet to identify themselves with the PHCC nurse at the beginning of every call they make as well as to login to the website. This will allow us to determine how many patients provided with the magnet call the PHCC/use the website as well as the number of times they call/login and their most common questions. The number on the magnet will allow us to determine of those who call/login to the PHCC, the number that complete the FOBT.

A four month follow-up patient survey will be conducted by the PHCC to evaluate patient experience with the PHCC and/or CRC Information and Screening Website as well as possible barriers to FOBT compliance. We will also conduct a survey of PCPs involved in the study to determine their experience with the study protocol and how to better facilitate PCP collaboration in research.

The study has been designed to be two-tailed with an alpha error of 0.05%, a beta error of 10% and a power index of 90%. Current FOBT screening rates in Manitoba are approximately 41.9% (Statistics Canada, 2009). It is believed that an intervention leading to an increase in FOBT screening rates of 15% would be clinically significant as it has been predicted that if approximately 70 % of Canadians aged 50 to 74 had a biennial FOBT, followed up by colonoscopy for positive FOBTs, the CRC mortality rate could be reduced by an estimated 17% (Statistics Canada, 2009). A logistic regression of a binary response variable (Y) on a binary independent variable (X) with a sample size of 716 observations [of which 80% are in the group that does not utilize the supplied intervention/magnet PHCC or Website (X=0) and 20% are in the group that does utilize the intervention/magnet PHCC or Website (X=1)] achieves 90% power at a 0.05 significance level to detect a change in Prob(Y=1) from the baseline value of 0.400 to 0.550. This change corresponds to an odds ratio of 1.833.

A biostatistician will be involved in the statistical analysis of results. Analysis of results will be based on the Intention to Treat Model. Therefore, patients not returning their FOBT test within a period of four months will be scored as failing to complete the FOBT test. Categorical variables will be compared using the Chi-square test or Fisher's exact test. The time taken to return FOBT cards will be estimated using Kaplan-Meier analysis. Statistical analysis will be performed using SAS or SPSS Software.

All forms provided to the PCP/Clinics will be collected by the study coordinator at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Average risk men and women
* between the ages of 50 to 74 years
* no symptoms of colorectal cancer
* no personal history of colorectal cancer, polyps or diseases of the colon requiring monitoring by colonoscopy
* includes individuals with one first degree relative with cancer of adenomatous polyps affected at age greater than 60 or two or more second degree relatives with polyps or cancer

Exclusion Criteria:

* walk-in patients
* patients having had a flexible sigmoidoscopy or double contrast barium enema within the last 5 years
* patients having had a colonoscopy within the last 10 years.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2395 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fecal Occult Blood Test (FOBT) completion rate | 4 months

SECONDARY OUTCOMES:
The most common patient questions and comments about colorectal cancer, screening, and the fecal occult blood test during the intervention(s). A patient and primary care provider survey. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alan Katz, MBChB, CCFP, MSc, Principal Investigator — University of Manitoba; Kathleen M Clouston, Ph.D., Study Director — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Clouston K, Katz A, Martens PJ, Sisler J, Turner D, Lobchuk M, McClement S, Crow G; CIHR/CCMB Team in Primary Care Oncology (PCO-NET). Does access to a colorectal cancer screening website and/or a nurse-managed telephone help line provided to patients by their family physician increase fecal occult blood test uptake?: results from a pragmatic cluster randomized controlled trial. BMC Cancer. 2014 Apr 16;14:263. doi: 10.1186/1471-2407-14-263. PMID 24739235
- [Derived] Clouston K, Katz A, Martens PJ, Sisler J, Turner D, Lobchuk M, McClement S; CIHR/CCMB Team in Primary Care Oncology (PCO-NET). Does access to a colorectal cancer screening website and/or a nurse-managed telephone help line provided to patients by their family physician increase fecal occult blood test uptake?: A pragmatic cluster randomized controlled trial study protocol. BMC Cancer. 2012 May 17;12:182. doi: 10.1186/1471-2407-12-182. PMID 22607726
- See also: BMC Cancer (Published Protocol) — http://www.biomedcentral.com/1471-2407/12/182